CLINICAL TRIAL: NCT03526172
Title: Assessing Physical Activity Levels of Patients Following High Tibial Osteotomy (HTO) With and Without Bone Grafting.
Brief Title: Assessing Physical Activity Levels of Patients Following HTO.
Status: Terminated | Type: Observational
Why Stopped: Halting of all research and elective surgeries due to the Covid-19 pandemic
Sponsor: University of Winchester (Other)
Collaborators: Hampshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: UMT057/13
Record Dates: First submitted 2018-04-21; First posted 2018-05-16 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: High Tibial Osteotomy With Allograft Wedge; High Tibial Osteotomy Without Allograft Wedge; Pre- and Post-operative Physical Activity Levels
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Patients undergoing HTO without the inclusion of any bone wedge
  Interventions: Procedure: High tibial osteotomy; Device: Accelerometer; Other: Questionnaire
- Allograft: Patients undergoing HTO with the inclusion of an allograft bone wedge
  Interventions: Procedure: High tibial osteotomy; Device: Allograft wedge; Device: Accelerometer; Other: Questionnaire

INTERVENTIONS:
Procedure: High tibial osteotomy — Uni-lateral medial opening-wedge high tibial osteotomy following a minimally invasive approach.
Device: Allograft wedge — Insertion of allograft wedge into the osteotomy gap during the HTO procedure
  Groups: Allograft
Device: Accelerometer — ActivPal accelerometer attached to thigh of patient to collect objective physical activity data at pre-determined intervals before and after surgery
Other: Questionnaire — Validated clinical questionnaires administered to patients to collect subjective physical activity data at pre-determined intervals before and after surgery

SUMMARY:
High tibial osteotomy (HTO is often indicated in physically active patients. The insertion of a bone graft during surgery has been shown to have good clinical and biomechanical outcomes, however objective data regarding post-surgery physical activity (PA) levels in patients who have undergone HTO with and without bone grafts does not exist in the literature.

Using accelerometers and questionnaires, this study will be the first to investigate this in an objective way.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing unilateral medial opening wedge high tibial osteotomy at Basingstoke & North Hampshire Hospital, UK

Exclusion Criteria:

* Concurrent procedures during HTO surgery
* The use of an off-loader knee brace in the 3 weeks leading up to surgery
* Revision surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective HTO patients on a patient database at Basingstoke & North Hampshire Hospital, UK.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Objective physical activity levels (measured in steps per day) | 14 weeks per patient
  Physical activity data (step-count and body position) collected via an accelermeter that is attached to the thigh for 7 day periods at pre-determined intervals before and after surgery
Intensity of physical activity (measured in steps per minute) | 14 weeks per patient
  Physical activity data (step-count and body position) collected via an accelermeter that is attached to the thigh for 7 day periods at pre-determined intervals before and after surgery

SECONDARY OUTCOMES:
Subjective reasons, thoughts and feelings behind post-operative physical activity levels (thematic analysis) | 1 hour per patient
  interviews with fully healed patients to determine their reasons, thoughts and feelings behind their post-operative levels of physical activity
Subjective physical activity levels | 14 weeks per patient
  Physical activity data (step-count and body position) collected via the implementation of validated questionnaires at pre-determined intervals before and after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Simon Jobson, Study Director — University of Winchester
Locations (1):
- University of Winchester, Winchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be made available to other researchers. Aggregated and analysed data will be anonymised and included in publications in peer-reviewed journals

REFERENCES:
- [Background] Copeland JL, Esliger DW. Accelerometer assessment of physical activity in active, healthy older adults. J Aging Phys Act. 2009 Jan;17(1):17-30. doi: 10.1123/japa.17.1.17. PMID 19299836
- [Background] Eisenberg MH, Phillips LA, Fowler L, Moore PJ. The Impact of E-diaries and Accelerometers on Young Adults' Perceived and Objectively Assessed Physical Activity. Psychol Sport Exerc. 2017 May;30:55-63. doi: 10.1016/j.psychsport.2017.01.008. Epub 2017 Jan 31. PMID 28966555
- [Background] Falck RS, Landry GJ, Brazendale K, Liu-Ambrose T. Measuring Physical Activity in Older Adults Using MotionWatch 8 Actigraphy: How Many Days are Needed? J Aging Phys Act. 2017 Jan;25(1):51-57. doi: 10.1123/japa.2015-0256. Epub 2016 Aug 24. PMID 27281368
- [Background] Martins RC, Reichert FF, Bielemann RM, Hallal PC. One-year Stability of Objectively Measured Physical Activity in Young Brazilian Adults. J Phys Act Health. 2017 Mar;14(3):208-212. doi: 10.1123/jpah.2015-0384. Epub 2016 Dec 20. PMID 27997276